# CASE REPORT FORM (CRF)

# CAD-EYE VS. White Light: A Multi-Centric Study **ELIGIBILITY FORM**

| Patient number: | | Date: | | | |
|---|---|---|---|---|---|
| Date of birth: | | Gender: | Fem | nale 🗌 | Male |
| Length (cm) | | Weight (kg) | | | |
| ı | NCLUSION CRITERIA | | | Yes | No |
| 1. Subject is 40-80 | years old | | | | |
| 2. Subject is under | going colonoscopy for | the following | | | |
| a. Primary CRO | Screening | | | | |
| b. Post-polype | ctomy surveillance | | | | |
| c. Work up fol | lowing FIT positivity | | | | |
| d. Symptoms/ | signs suspicions of CRC | | | | |
| 3. Subjects must be willing to give written informed consent for | | | | | |

| EXCLUSION CRITERIA | YES | No |
|------------------------------------------|-----|----|
| 1. Patient is: <40 years old | | |
| 2. Unable to consent | | |
| 3. Contraindicated to undergo endoscopy, | | |

the trial

| 4. Already hospitalized for another illness |
|-----------------------------------------------------|
| 5. Pregnant or lactating |
| 6. Patients with the following conditions: |
| History of colon resection |
| History of CRC |
| Antithrombotic therapy precluding colon resection |
| Inflammatory Bowel Disease (IBD) |
| Familial Adenomatous Polyposis (FAP) |
| 7. Poor bowel preparation: BBPS 0 or 1 in a segment |
| RANDOMIZATION |
| White-light |
| CAD-EYE |
| INFORMED CONSENT SIGNED: |
| YES |
| □NO |
| Date consented: |

| PATIENT INFO |
|---------------------------------|
| Date & time of admission: |
| Indication for colonoscopy: |
| Surveillance |
| GI Symptoms, please specify: |
| Per-rectal bleeding |
| Abdominal pain |
| Weight loss |
| Primary CRC Screening |
| Family history of CRC |
| FIT positive |
| Other: |
| Drug History: |
| Anti-thrombotics. If yes, dose: |
| Others: |
| 1. |
| 2. |
| 3. |
| 4. |
| 5. |

| Endoscopic History: | |
|----------------------------------------------------|-------|
| No previous history | |
| Previous endoscopy (please list summary of report) | |
| 1. | Date: |
| 2. | Date: |
| 3. | Date: |
| 4. | Date: |

| PROCEDURAL INFO |
|------------------------------------------------------------|
| Endoscopy: |
| Date of procedure: |
| Endoscope system used: |
| Intubation: Yes No |
| Propofol: Yes, mention dosage mg |
| □No |
| Midazolam: Yes, mention dosage mg |
| □No |
| Blood pressure: (mmHg) |
| O2 saturation: % |
| Pulse: (b/m) |
| BBPS Score (0-9) |
| Right colon: |
| Transverse colon: |
| Left colon: |
| Intraprocedural information: |
| Insertion time (min): |
| Withdrawal time (min): |
| Ileocecal valve intubation: yes/ no |
| If yes, please provide time: Min |
| if no, please specify distance from anal verge reached: cm |

| Post procedural Information: |
|------------------------------------------------------|
| Patient Excluded from study (post procedure): Yes No |
| If yes, please provide reason: |
| Adverse Events |
| None |
| GI Symptoms |
| Perforation |
| Hemorrhage |
| Infection |
| Others: |

## WHITE LIGHT FORM

| Poly <sub> </sub> | olyps (Number) • Lesion |
|-------------------|-------------------------------------------------|
| • | Container |
| • | Site location |
| | o Segment: |
| | ■ Rectum |
| | ■ Sigmoid |
| | ■ Left colon |
| | ■ Transverse colon |
| | ■ Right colon |
| | ■ Cecum |
| | <ul><li>Distance from anal verge (cm)</li></ul> |
| • | Paris type (check appendix): |
| | ○ □0-1p |
| | ○ □0-1ps |
| | ○ <b>0-1</b> s |
| | ○ □0-IIa |
| | o O-IIb |
| | ○ □0-IIc |
| | o |
| • | Polypectomy: |
| | ○ YES: |
| | ○ □NO: |

| • | Biopsy for histopathology: |
|---|-----------------------------------------------------------------|
| | ○ YES: |
| | o |
| • | Histopathology result: |
| | <ul> <li>Hyperplastic</li> </ul> |
| | Adenoma with no dysplasia |
| | Adenoma with low grade dysplasia |
| | Adenoma with high grade dysplasia |
| | Adenocarcinoma in situ |
| | <ul> <li>Adenocarcinoma</li> </ul> |
| | o Others: |
| • | Characterization (white light Endoscopic assessment of lesion): |
| | <ul> <li>Hyperplastic</li> </ul> |
| | o Adenoma |
| • | Characterization (BLI Endoscopic assessment of lesion): |
| | ○ Hyperplastic |
| | o Adenoma |
| • | Images for each polyp: |
| | ○ <b>Yes</b> |
| | ○ |
| • | Remarks: |

## **CAD-EYE FORM**

| POLYP (Number) |
|-------------------------------------------------|
| • Lesion |
| Container |
| Site location |
| <ul> <li>Segment</li> </ul> |
| ■ Rectum |
| ■ Sigmoid |
| ■ Left colon |
| ■ Transverse colon |
| ■ Right colon |
| ■ Cecum |
| <ul><li>Distance from anal verge (cm)</li></ul> |
| <ul><li>Paris type (check appendix):</li></ul> |
| o 0-1p |
| o 0-1ps |
| o 0-1s |
| o 0-IIa |
| o 0-IIb |
| o 0-IIc |
| o |
| <ul> <li>Polypectomy</li> </ul> |
| ○ |

| | $\circ$ $\square$ NO |
|---|-----------------------------------------------------------------|
| • | Biopsy for histopathology |
| | ○ <b>YES</b> |
| | o |
| • | Histopathology result: |
| | <ul> <li>Hyperplastic</li> </ul> |
| | <ul> <li>Hyperplastic</li> </ul> |
| | Adenoma with no dysplasia |
| | Adenoma with low grade dysplasia |
| | <ul> <li>Adenoma with high grade dysplasia</li> </ul> |
| | Adenocarcinoma in situ |
| | <ul> <li>Adenocarcinoma</li> </ul> |
| | o Others: |
| • | Characterization (white light Endoscopic assessment of lesion): |
| | <ul> <li>Hyperplastic</li> </ul> |
| | o Adenoma |
| • | Characterization (BLI Endoscopic assessment of lesion): |
| | <ul> <li>Hyperplastic</li> </ul> |
| | o Adenoma |
| • | CAD EYE Detection of lesion |
| | ○ Yes: |
| | o |
| • | Characterization (by CAD-EYE): |
| | <ul> <li>Hyperplastic</li> </ul> |

| | <ul> <li>Adenoma</li> </ul> |
|---|--------------------------------------------------------------------------|
| • | CAD EYE Accuracy of lesion |
| | ○ <b>FN</b> |
| | ○ □TP-C |
| | o ПТР-Е |
| | ○ <b>FP</b> |
| • | IN CASE of resection: |
| | <ul> <li>CAD Characterization of resection plane</li> </ul> |
| | <ul> <li>CAD eye detected residual lesions at resection edges</li> </ul> |
| | • Yes |
| | • |
| | <ul> <li>If yes what was your next step:</li> </ul> |
| | <ul> <li>Took another biopsy from edges</li> </ul> |
| | <ul> <li>More resection of the residual lesions</li> </ul> |
| | <ul> <li>No further action</li> </ul> |
| • | Images for each polyp |
| | ○ Yes |
| | <ul><li>○ No</li></ul> |
| • | Remarks: |

#### **Appendix**

#### **Paris classification:**

1) Polypoid:

0-1p: pedunculated

0-1ps: Subpendunculated

0-1s: Sessile polyps2) Non-polypoid lesions:

0-IIa: superficial slightly elevated

0-IIb: flat

0-IIc: superficial depressed

0-III: excavated

#### **CAD EYE Accuracy of Lesion**

| | Endoscopist | CAD EYE |
|----------------------|------------------------|--------------------|
| False Negative (FN) | Detected | Not Detected |
| | And | |
| | Confirmed as Polyp | |
| False Positive (FP) | Not Detected | Detected |
| , , | And | |
| | Confirmed as Not Polyp | |
| True Positive CADEYE | Not Detected | Detected |
| (TP-C) | Before | And |
| (11 3) | CAD Eye alarm | Confirmed as Polyp |
| True Positive | Detected | Detected |
| Endoscopist (TP-E) | And | And |
| | Confirmed as Polyp | Confirmed as Polyp |